CLINICAL TRIAL: NCT06899035
Title: Evaluation of the Effects of Hydrotherapy on Balance and Selective Motor Control in Children With Cerebral Palsy
Brief Title: Effects of Hydrotherapy in Children With Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Melis Gökçe Dağbağ, Medical Doctor, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREH-FTR-MGDS-001
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy Children
Keywords: hydrotherapy; rehabilitation; balance; selective motor control; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: two groups: an intervention group and a control group
Who Masked: Outcomes Assessor
Masking Description: This is a single blind study, the control group will receive a home exercise program, while the intervention group will receive both a home exercise program and hydrotherapy. Outcome assessments will be conducted by an investigator who is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in the study group will undergo individualized water-based exercises (including standing, balance, weight shifting, breathing exercises, range of motion, stretching, and strengthening exercises) under the supervision of an experienced physiotherapist, 2-3 times per week for six weeks. Additionally, routine conventional exercises will be continued daily for six weeks.
  Interventions: Other: Intervention Group (water-based and conventional exercise)
- Control Group (Active Comparator): Patients in the control group will continue passive, active, active-assisted, or resistance-based upper and lower extremity conventional exercises appropriate to their functional level and muscle strength. They will be instructed to perform these exercises 2-3 times per week, with each session lasting no more than 45 minutes, for six weeks.
  Interventions: Other: control group (conventional exercise)

INTERVENTIONS:
Other: Intervention Group (water-based and conventional exercise) — Patients in the study group will undergo individualized water-based exercises (including standing, balance, weight shifting, breathing exercises, range of motion, stretching, and strengthening exercises) under the supervision of an experienced physiotherapist, 2-3 times per week for six weeks. Additionally, routine conventional exercises will be continued daily for six weeks.
  Arms: Intervention Group
Other: control group (conventional exercise) — Patients in the control group will continue passive, active, active-assisted, or resistance-based upper and lower extremity conventional exercises appropriate to their functional level and muscle strength. They will be instructed to perform these exercises 2-3 times per week, with each session lasting no more than 45 minutes, for six weeks.
  Arms: Control Group

SUMMARY:
The goal of this observational study is to learn the effects of hydrotherapy in children with cerebral palsy. It aims to answer if hydrotherapy is affective on balance and selective motor control of the children with cerebral palsy.

DETAILED DESCRIPTION:
Children diagnosed with cerebral palsy by a pediatric neurologist and followed up at the Pediatric Rehabilitation Outpatient Clinic of the Physical Medicine and Rehabilitation Department at Sağlık Bilimleri University Gaziosmanpaşa Training and Research Hospital, aged between 4 and 18 years, with a Gross Motor Function Classification System (GMFCS) level of 1-4, will be included in the study.

Patients scheduled for hydrotherapy treatment will be enrolled in the study. The participants will be randomly assigned into two groups using the envelope randomization method. The first group will be the study group, while the second group will be the control group. The control group will receive hydrotherapy after the study is completed.

Demographic data such as age, height, weight, and body mass index (BMI) of the included children will be recorded. Functional status will be assessed using the Gross Motor Function Classification System (GMFCS) and the Gross Motor Function Measure (GMFM-88) sections D and E. Balance will be evaluated with the Pediatric Balance Scale (PBS), selective motor control for upper and lower extremities with SCUES (Selective Control of Upper Extremity Scale) and SCALE (Selective Control Assessment of the Lower Extremity), activity with the Pediatric Functional Independence Measure (WeeFIM), participation with the Child and Adolescent Scale of Participation (CASP), quality of life with the Pediatric Quality of Life Inventory (PedsQL), and goal achievement with the Goal Attainment Scale (GAS).

Patients in the study group will undergo individualized water-based exercises (including standing, balance, weight shifting, breathing exercises, range of motion, stretching, and strengthening exercises) under the supervision of an experienced physiotherapist, 2-3 times per week for six weeks. Additionally, routine conventional exercises will be continued daily for six weeks.

Patients in the control group will continue passive, active, active-assisted, or resistance-based upper and lower extremity conventional exercises appropriate to their functional level and muscle strength. They will be instructed to perform these exercises 2-3 times per week, with each session lasting no more than 45 minutes, for six weeks.

Assessments conducted at the beginning of the study will be repeated at the end of six weeks and one month after the completion of the intervention. The results will be compared accordingly.

* Conventional exercise therapy consists of range of motion, stretching, and strengthening exercises applied to patients diagnosed with cerebral palsy.

This is a single-center, single-blind, prospective clinical study. A total of 36 patients, including 18 in the study group and 18 in the control group, are planned to be included between January 1, 2024, and September 15, 2025.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Cerebral Palsy by a specialist physician
* Aged between 4-18 years
* Cooperative with physiotherapy applications
* Gross Motor Function Classification System (GMFCS) levels 1-4
* Willing to participate in the study and undergo assessments

Exclusion Criteria:

* Mental retardation or insufficient cognitive function to comply with study assessments
* GMFCS level 5
* Presence of an intrathecal baclofen pump for spasticity treatment or history of soft tissue and/or bone surgery
* Active infection or localized skin infection at the injection site
* History of active seizures
* Presence of contractures
* Serious systemic disease that may prevent exercise participation
* Injury and/or surgery within the last 6 months
* Botulinum toxin injection within the last 6 months
* Contraindications to hydrotherapy, including severe fear of water, behavioral problems, shortness of breath at rest, infection, incontinence, known chlorine allergy, open wounds, acute systemic illness, epilepsy, tracheostomy, permanent drains, immunodeficiency.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Pediatric Balance Scale | six weeks
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills during tasks that mimic experiences of everyday living in school-aged children. The scale consists of 14 balance-related test items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.

SECONDARY OUTCOMES:
Selective Control of Upper Extremity Scale (SCUES) | six weeks
  Selective Control of Upper Extremity Scale is a clinical assessment tool used to evaluate selective motor control (SMC) in the upper extremities of individuals with neurological impairments, such as cerebral palsy. It is adapted from the Selective Control Assessment of the Lower Extremity (SCALE) and focuses on assessing isolated joint movements in the shoulder, elbow, forearm, wrist, and fingers while minimizing synergistic patterns or involuntary movements.
Selective Control Assessment of the Lower Extremity (SCALE) | six weeks
  Selective Control Assessment of the Lower Extremity is a clinical tool used to evaluate selective voluntary motor control (SVMC) in individuals with neuromotor disorders, such as cerebral palsy. It assesses the ability to perform isolated joint movements in the lower extremities without involuntary movements or abnormal muscle synergies.

OTHER OUTCOMES:
Goal Attainment Scaling (GAS) | six weeks
  Goal Attainment Scaling is a method of scoring the extent to which patient's individual goals are achieved in the course of intervention. In effect, each patient has their own outcome measure but this is scored in a standardised way as to allow statistical analysis.
Pediatric Quality of Life Inventory (PedsQL). | six weeks
  Pediatric Quality of Life Inventory is a standardized tool designed to measure health-related quality of life (HRQoL) in children and adolescents. It assesses the physical, emotional, social, and school functioning of children with various health conditions, including cerebral palsy.
Child and Adolescent Scale of Participation (CASP). | six weeks
  Child and Adolescent Scale of Participation is a standardized assessment tool used to measure the extent of participation of children and adolescents in daily life activities across various settings, such as home, school, and community. It is particularly useful for children with disabilities or developmental disorders, including cerebral palsy.
Pediatric Functional Independence Measure (WeeFIM) | six weeks
  Pediatric Functional Independence Measure is a standardized tool used to assess functional independence in children with disabilities, including cerebral palsy. It evaluates a child's ability to perform daily activities and tracks their level of assistance required in different domains.
Gross Motor Function Classification System (GMFCS) | six weeks
  The Gross Motor Function Classification System is a standardized tool used to classify gross motor function in children and adolescents with cerebral palsy. It categorizes mobility levels based on self-initiated movement, need for assistive devices, and functional limitations.
Gross Motor Function Measure (GMFM-88) | six weeks
  The Gross Motor Function Measure is a standardized clinical tool used to assess gross motor function in children with cerebral palsy and other motor impairments. It evaluates changes in motor abilities over time and helps guide rehabilitation planning.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Yılmaz Yalçınkaya, Study Director — Gaziosmanpasa Research and Education Hospital
Locations (1):
- GaziosmanpasaTREH, Istanbul, Gaziosmanpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roostaei M, Baharlouei H, Azadi H, Fragala-Pinkham MA. Effects of Aquatic Intervention on Gross Motor Skills in Children with Cerebral Palsy: A Systematic Review. Phys Occup Ther Pediatr. 2017 Oct 20;37(5):496-515. doi: 10.1080/01942638.2016.1247938. Epub 2016 Dec 14. PMID 27967298
- [Background] Retarekar R, Fragala-Pinkham MA, Townsend EL. Effects of aquatic aerobic exercise for a child with cerebral palsy: single-subject design. Pediatr Phys Ther. 2009 Winter;21(4):336-44. doi: 10.1097/PEP.0b013e3181beb039. PMID 19923974